CLINICAL TRIAL: NCT05878873
Title: The Neural Underpinnings and the Impact of Wearable Sensory Stimulation During Split-belt Treadmill Adaptation in People With Multiple Sclerosis
Brief Title: The Neural Mechanisms of Split-belt Treadmill Adaptation in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Brett Fling, Associate Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1664
Record Dates: First submitted 2023-05-12; First posted 2023-05-26 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: split-belt treadmill; adaptation; multiple sclerosis; functional near-infrared spectroscopy; cortical activation; gait asymmetry; locomotion; sensorimotor control
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Split-belt Treadmill Training without TENS (Sham Comparator): During this arm, participants will perform split-belt treadmill training with sensory stimulation equipment outfitted but not active during all adaptation sessions.
  Interventions: Behavioral: Split-belt Treadmill
- Split-belt Treadmill Training with TENS (Experimental): During this arm, participants will perform split-belt treadmill training with active sensory stimulation occuring simultaneously during all adaptation sessions.
  Interventions: Behavioral: Split-belt Treadmill; Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Behavioral: Split-belt Treadmill — Split-belt treadmill training, where the speed of each leg is controlled independently has been shown to create gait adaptation where the coordination of each leg is altered, creating improved gait symmetry for people with walking impairments.
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS is a form of nerve stimulation that stimulates at a frequency below motor threshold, targeting activation of sensory receptors, such as muscle spindles. Electrodes that create this stimulation will be placed on the skin superficial to the muscle bellies of the tibialis anterior and rectus femoris.
  Arms: Split-belt Treadmill Training with TENS

SUMMARY:
Majority of people with multiple sclerosis experience difficulty with balance and mobility, leading to an increased risk of falls. The goal of this clinical trial is to learn about brain activity during walking adaptation in people with multiple sclerosis. Also, this clinical trial will test a form of nerve stimulation to see if it can improve walking performance.

The main questions it aims to answer are:

* What areas of the brain are the most active during walking adaptation?
* Can nerve stimulation make walking adaptation more effective?

Participants will walk on a treadmill where each leg will go a different speed which will create walking adaptation. At the same time, brain scans will occur. There will be two sessions of walking adaptation, one with nerve stimulation, and one without nerve stimulation. Researchers will compare people with multiple sclerosis to healthy young adults to see if there are differences in brain activity.

DETAILED DESCRIPTION:
Most people with MS (PwMS) experience significant gait asymmetries between the two legs leading to an increased risk of falls and musculoskeletal injury. The objective of this study is to investigate the neural mechanisms of gait adaptation and the effects of transcutaneous electrical nerve stimulation (TENS) on adaptability during split-belt treadmill training in PwMS. Our hypothesis is that TENS will strengthen sensorimotor integration via amplified afferent signaling, thereby enhancing adaptation, and further improving gait symmetry chronically. Functional near-infrared spectroscopy (fNIRS) will be used during a split-belt treadmill training paradigm to assess cortical activation during gait adaptation. Additionally, the effect of split-belt treadmill training coupled with TENS on gait adaptability in PwMS will be tested with experimental and a sham TENS split-belt treadmill sessions. Cortical activation and the effect of TENS on gait adaptability will be compared between young neurotypical adults and PwMS to assess differences that can be attributed to multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of relapsing remitting multiple sclerosis OR a neurotypical adult (ages 18-86)
* Not experiencing an active relapse
* Able to stand and walk without an assistive device
* Able to walk for three tenths of a mile without stopping to rest

Exclusion Criteria:

* Unable to walk for three tenths of a mile without assistance
* Musculoskeletal injury in past 6 months
* Lower extremity surgery in past 6 months
* Unable to abstain from medications that impair balance
* Currently pregnant
* History of traumatic brain injury
* History of vestibular disease
* History of any other balance impairment unrelated to multiple sclerosis

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett W Fling, Ph.D., Principal Investigator — Colorado State University
Locations (1):
- The Sensorimotor Neuroimaging Laboratory, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The data will not publicly available due to participant privacy.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 55 participants consented to be screened for eligibility, and 51 participants (31 people with multiple sclerosis and 20 healthy controls) were enrolled.
Groups:
- Split-belt Treadmill Training With TENS First: During this arm, participants will perform split-belt treadmill training with sensory stimulation equipment outfitted and active for the first training session but not active during the second session.
- Split-belt Treadmill Training With TENS Second: During this arm, participants will perform split-belt treadmill training with active sensory stimulation equipment outfitted but not active during the first training session, and active during the second training session.
Period: Overall Study
Arm/Group | Split-belt Treadmill Training With TENS First | Split-belt Treadmill Training With TENS Second
Started | 24 | 27
People With Multiple Sclerosis Started: | 15 | 16
People With Multiple Sclerosis Completed: | 13 | 16
Healthy Controls Started: | 9 | 11
Healthy Controls Completed: | 9 | 11
Completed | 22 | 27
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: This population contained 28 people with multiple sclerosis and 20 healthy controls.
Groups:
- Total: Total of all reporting groups
Arm/Group | Split-belt Treadmill Training With TENS First | Split-belt Treadmill Training With TENS Second | Total
Number analyzed (Participants) | 22 | 26 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Rows are split between people with multiple sclerosis and healthy controls.
  years
    People with Multiple Sclerosis: number analyzed (Participants) | 13 | 15 | 28
    People with Multiple Sclerosis | 55.5 (9.1) | 52.2 (11.6) | 53.7 (10.5)
    Healthy Controls: number analyzed (Participants) | 9 | 11 | 20
    Healthy Controls | 57.3 (11.9) | 50.9 (15.5) | 53.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Rows are split between people with multiple sclerosis and healthy controls.
  Participants
    People with Multiple Sclerosis: number analyzed (Participants) | 13 | 15 | 28
    People with Multiple Sclerosis: Female | 8 | 11 | 19
    People with Multiple Sclerosis: Male | 5 | 4 | 9
    Healthy Controls: number analyzed (Participants) | 9 | 11 | 20
    Healthy Controls: Female | 6 | 6 | 12
    Healthy Controls: Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Rows are split between people with multiple sclerosis and healthy controls.
  Participants
    People with Multiple Sclerosis: number analyzed (Participants) | 13 | 15 | 28
    People with Multiple Sclerosis: Hispanic or Latino | 1 | 0 | 1
    People with Multiple Sclerosis: Not Hispanic or Latino | 12 | 15 | 27
    People with Multiple Sclerosis: Unknown or Not Reported | 0 | 0 | 0
    Healthy Controls: number analyzed (Participants) | 9 | 11 | 20
    Healthy Controls: Hispanic or Latino | 0 | 0 | 0
    Healthy Controls: Not Hispanic or Latino | 9 | 11 | 20
    Healthy Controls: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Rows are split between people with multiple sclerosis and healthy controls.
  Participants
    People with Multiple Sclerosis: number analyzed (Participants) | 13 | 15 | 28
    People with Multiple Sclerosis: American Indian or Alaska Native | 0 | 0 | 0
    People with Multiple Sclerosis: Asian | 0 | 0 | 0
    People with Multiple Sclerosis: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    People with Multiple Sclerosis: Black or African American | 0 | 1 | 1
    People with Multiple Sclerosis: White | 13 | 14 | 27
    People with Multiple Sclerosis: More than one race | 0 | 0 | 0
    People with Multiple Sclerosis: Unknown or Not Reported | 0 | 0 | 0
    Healthy Controls: number analyzed (Participants) | 9 | 11 | 20
    Healthy Controls: American Indian or Alaska Native | 0 | 0 | 0
    Healthy Controls: Asian | 0 | 0 | 0
    Healthy Controls: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Healthy Controls: Black or African American | 0 | 0 | 0
    Healthy Controls: White | 9 | 11 | 20
    Healthy Controls: More than one race | 0 | 0 | 0
    Healthy Controls: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Cortical Activation
Description: Cortical activation is measured using functional near-infrared spectroscopy (fNIRS) during split-belt treadmill walking. Hemodynamic responses are modeled using a general linear model (GLM) applied to the oxyhemoglobin (HbO) signal. The model includes regressors for distinct phases of walking, with the primary contrast comparing early adaptation (strides 6-30 after split-belt onset) to a baseline walking period. The outcome is defined as the difference in this HbO beta weight contrast with TENS ON compared to TENS OFF. Activation is averaged across all fNIRS channels to provide a whole-brain estimate of cortical activity. A larger value indicates a greater increase in activation from baseline walking to early adaptation. This was measured on both training session 1 and training session 2 to account for the crossover design (i.e. participants are receiving TENS on different days).
Time Frame: Training session 1 (day 1), training session 2 (day 28)
Population: The sample included 28 individuals with multiple sclerosis and 20 healthy controls. A randomized crossover design was used, with each participant receiving TENS ON during one training session and TENS OFF during the other.
Measure: Least Squares Mean (Standard Error); unit: Unitless GLM beta weight (HbO)
Groups:
- Split-belt Treadmill Training Without TENS: During this arm, participants will perform split-belt treadmill training with sensory stimulation equipment outfitted but not active during adaptation.
  Split-belt Treadmill: Split-belt treadmill training, where the speed of each leg is controlled independently has been shown to create gait adaptation where the coordination of each leg is altered, creating improved gait symmetry for people with walking impairments.
- Split-belt Treadmill Training With TENS: During this arm, participants will perform split-belt treadmill training with active sensory stimulation occuring simultaneously during adaptation.
  Split-belt Treadmill: Split-belt treadmill training, where the speed of each leg is controlled independently has been shown to create gait adaptation where the coordination of each leg is altered, creating improved gait symmetry for people with walking impairments.
  Transcutaneous Electrical Nerve Stimulation (TENS): TENS is a form of nerve stimulation that stimulates at a frequency below motor threshold, targeting activation of sensory receptors, such as muscle spindles. Electrodes that create this stimulation will be placed on the skin superficial to the muscle bellies of the tibialis anterior and rectus femoris.
Arm/Group | Split-belt Treadmill Training Without TENS | Split-belt Treadmill Training With TENS
Number analyzed (Participants) | 48 | 48
Unitless GLM beta weight (HbO)
  People with Multiple Sclerosis: number analyzed (Participants) | 28 | 28
  People with Multiple Sclerosis | 0.054 (0.021) | -0.024 (0.021)
  Healthy Controls: number analyzed (Participants) | 20 | 20
  Healthy Controls | 0.074 (0.025) | -0.016 (0.025)
Statistical Analysis 1: Comparison: Split-belt Treadmill Training Without TENS vs Split-belt Treadmill Training With TENS; Statistical analysis comparing cortical activation between TENS ON and TENS OFF conditions in people with multiple sclerosis; Test type: Other; p = 0.007, Mixed Models Analysis — This value was adjusted using false discovery rate; Degrees of freedom = 44; Mean Difference (Net) = -0.078, Standard Error of Mean 0.027 — This estimate calculation is TENS ON - TENS OFF
Statistical Analysis 2: Comparison: Split-belt Treadmill Training Without TENS vs Split-belt Treadmill Training With TENS; Statistical analysis comparing cortical activation between TENS ON and TENS OFF conditions in healthy controls; Test type: Other; p = 0.008, Mixed Models Analysis — This value was adjusted using false discovery rate; Degrees of freedom = 44; Mean Difference (Net) = -0.089, Standard Error of Mean 0.032 — The estimate calculation is TENS ON - TENS OFF

2. Primary Outcome: Change in Adaptation Savings
Description: Adaptation savings is defined as the difference in early adaptation performance between training session 1 (Day 1) and training session 2 (Day 28) during split-belt treadmill walking. Early adaptation is quantified using relative step length asymmetry (SLA), calculated from strides 6 to 30 following split-belt onset. SLA is computed from three-dimensional motion capture and force data as the difference between step lengths of the legs, normalized to total stride length:
  SLA = (Step Length_fast - Step Length_slow) / (Step Length_fast + Step Length_slow).
  This yields a unitless measure of asymmetry. The outcome measure is the difference in SLA between visits (training session 2 - training session 1). Larger values reflect faster adaptation at training session 2, consistent with retention of prior learning.
Time Frame: Training session 1 (day 1), training session 2 (day 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Unitless Relative Step Length Asymmetry
Arm/Group | Split-belt Treadmill Training With TENS First | Split-belt Treadmill Training With TENS Second
Number analyzed (Participants) | 22 | 26
Unitless Relative Step Length Asymmetry
  People with Multiple Sclerosis: number analyzed (Participants) | 13 | 15
  People with Multiple Sclerosis | 0.0032 (0.0103) | 0.0451 (0.0096)
  Healthy Controls: number analyzed (Participants) | 9 | 11
  Healthy Controls | 0.0221 (0.0124) | 0.0278 (0.0112)
Statistical Analysis 1: Comparison: Split-belt Treadmill Training With TENS First vs Split-belt Treadmill Training With TENS Second; Statistical analysis comparing savings between TENS ON and TENS OFF conditions in people with multiple sclerosis; Test type: Other; p = 0.014, Mixed Models Analysis — This value was adjusted using false discovery rate; Degrees of freedom = 44; Mean Difference (Net) = 0.0420, Standard Error of Mean 0.0141 — This estimate calculation is TENS ON - TENS OFF at Visit 2
Statistical Analysis 2: Comparison: Split-belt Treadmill Training With TENS First vs Split-belt Treadmill Training With TENS Second; Statistical analysis comparing savings between TENS ON and TENS OFF conditions in healthy controls; Test type: Other; p = 0.878, Mixed Models Analysis — This value was corrected with false discovery rate; Degrees of freedom = 44; Mean Difference (Net) = -0.0058, Standard Error of Mean 0.167 — The estimate calculation is TENS ON - TENS OFF at Visit 2

3. Primary Outcome: Rate of Step Length Asymmetry Adaptation
Description: Step length asymmetry during early adaptation, representing the rate of adaptation. Early adaptation is quantified using relative step length asymmetry (SLA), calculated from strides 6 to 30 following split-belt onset. SLA is computed from three-dimensional motion capture and force data as the difference between step lengths of the legs, normalized to total stride length:
  SLA = (Step Length_fast - Step Length_slow) / (Step Length_fast + Step Length_slow).
  This yields a unitless measure of asymmetry. The outcome measure is the difference in early adaptation SLA during TENS ON compared to TENS OFF. Values closer to zero reflect faster adaptation.This analysis was performed only on data from each participant's first visit to avoid known effects of increased adaptation rate (learning) during subsequent exposures.
Time Frame: Training session 1 (day 1)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Unitless Relative Step Length Asymmetry
Arm/Group | Split-belt Treadmill Training Without TENS | Split-belt Treadmill Training With TENS
Number analyzed (Participants) | 26 | 22
Unitless Relative Step Length Asymmetry
  People with Multiple Sclerosis: number analyzed (Participants) | 15 | 13
  People with Multiple Sclerosis | -0.090 (0.012) | -0.088 (0.013)
  Healthy Controls: number analyzed (Participants) | 11 | 9
  Healthy Controls | -0.095 (0.014) | -0.103 (0.016)
Statistical Analysis 1: Comparison: Split-belt Treadmill Training Without TENS vs Split-belt Treadmill Training With TENS; Statistical analysis comparing rate of adaptation between TENS ON and TENS OFF conditions in people with multiple sclerosis; Test type: Other; p = 0.898, Mixed Models Analysis — This value was corrected using false discovery rate; Degrees of freedom = 44; Mean Difference (Final Values) = 0.002, Standard Error of Mean 0.018 — The estimate calculation is TENS ON - TENS OFF
Statistical Analysis 2: Comparison: Split-belt Treadmill Training Without TENS vs Split-belt Treadmill Training With TENS; Statistical analysis comparing rate of adaptation between TENS ON and TENS OFF conditions in healthy controls; Test type: Other; p = 0.698, Mixed Models Analysis — This value was corrected using false discovery rate; Degrees of freedom = 44; Mean Difference (Final Values) = -0.008, Standard Error of Mean 0.021 — The estimate calculation is TENS ON - TENS OFF

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during each study visit (visit 1 at day 1 and visit 2 at day 28) and between visits. Participants were not followed after study completion.
Description: Adverse event data were collected through participant self-report and investigator observation during each study visit. No adverse events occurred. Definitions of adverse and serious adverse events followed ClinicalTrials.gov guidance. No alternative definitions were used.
Groups:
- Split-belt Treadmill Training With TENS: People With Multiple Sclerosis: During this arm, participants with multiple sclerosis will perform split-belt treadmill training with active sensory stimulation occuring simultaneously during adaptation.
  Split-belt Treadmill: Split-belt treadmill training, where the speed of each leg is controlled independently has been shown to create gait adaptation where the coordination of each leg is altered, creating improved gait symmetry for people with walking impairments.
- Split-belt Treadmill Training Without TENS: People With Multiple Sclerosis: During this arm, participants with multiple sclerosis will perform split-belt treadmill training with sensory stimulation equipment outfitted but not active during adaptation.
  Split-belt Treadmill: Split-belt treadmill training, where the speed of each leg is controlled independently has been shown to create gait adaptation where the coordination of each leg is altered, creating improved gait symmetry for people with walking impairments.
- Split-belt Treadmill Training With TENS: Healthy Controls: During this arm, healthy control participants will perform split-belt treadmill training with active sensory stimulation occuring simultaneously during adaptation.
  Split-belt Treadmill: Split-belt treadmill training, where the speed of each leg is controlled independently has been shown to create gait adaptation where the coordination of each leg is altered, creating improved gait symmetry for people with walking impairments.
- Split-belt Treadmill Training Without TENS: Healthy Controls: During this arm, healthy control participants will perform split-belt treadmill training with sensory stimulation equipment outfitted but not active during adaptation.
  Split-belt Treadmill: Split-belt treadmill training, where the speed of each leg is controlled independently has been shown to create gait adaptation where the coordination of each leg is altered, creating improved gait symmetry for people with walking impairments.
Arm/Group | Split-belt Treadmill Training With TENS: People With Multiple Sclerosis | Split-belt Treadmill Training Without TENS: People With Multiple Sclerosis | Split-belt Treadmill Training With TENS: Healthy Controls | Split-belt Treadmill Training Without TENS: Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT05878873/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT05878873/ICF_001.pdf